CLINICAL TRIAL: NCT00515489
Title: Aggressiveness and Agitation of Acute Psychotic Patients: Influence in Safety and Effectiveness of Risperidone Treatment
Brief Title: Study on the Safety and Effectiveness of Risperidone Treatment of Acute Psychotic Patients
Status: Terminated | Type: Observational
Why Stopped: Due to the achievement of minimum required sample size and new changes in local regulations.
Sponsor: Janssen-Cilag, S.A. (Industry)
Responsible Party: Country Medical Director, Janssen-Cilag S.A., Spain
Other Study IDs: CR009214
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
Keywords: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 001: Risperidone as prescribed
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — as prescribed

SUMMARY:
The purpose of this study was to evaluate the safety of risperidone treatment in acute psychotic patients that require an admission into emergency department. The effectiveness of risperidone in controlling acute psychotic symptomatology and incidence, severity and risk of psychomotor agitation in acute psychotic patients was also studied.

DETAILED DESCRIPTION:
Antipsychotic drugs are key treatment for the acute psychotic symptoms experienced by schizophrenic, schizoaffective disorder and schizophreniform disorder patients. In the last years, atypical antipsychotics having fewer side effects than conventional neuroleptics, have been introduced into clinical practice. There is not an agreement about what type of drugs should be used in an emergency situation (acute psychotic patient). The aim of this observational, prospective study was to evaluate the impact of a treatment regimen with the atypical antipsychotic drug, risperidone, as first line treatment in acute psychotic patients that requested an admission into the hospital. Effectiveness of risperidone treatment was measured by Positive and Negative Syndrome Scale (PANSS) agitation sub scale, Brief Psychotic Rating Scale and days of in-patient period. Aggressive behavior was rated using Staff Observation Aggression Scale (SOAS) and Visual Analogic Scale for agitation and anxiety. Safety was evaluated collecting elicited adverse events. Observational study - Risperidone, 3-6 mg per day, orally, during the study period (in-patient period for each patient).

ELIGIBILITY:
Inclusion Criteria:

* Acute Psychotic symptoms in Schizophrenia
* Schizoaffective disorder and Schizophreniform disorders in patients that required an admission into a hospital and in which physicians considered the use of risperidone as treatment under clinical practice

Exclusion Criteria:

* Pregnant or lactating patients
* Patients with psychiatry pathology other than Schizophrenia or schizoaffective disorder
* Patients with neurology pathology except Parkinsonism induced by neuroleptics
* Patients with other severe concomitant pathology
* Patients treated with risperidone in the last 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Psychotic symptoms in Schizophrenia; Schizoaffective disorder and Schizophreniform disorders in patients that required an admission into a hospital and in which physicians considered the use of risperidone as treatment under clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 1882 (Actual)
Dates: Start 2001-11; Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Safety of risperidone treatment in acute psychotic patients that require an admission into emergency. | 3 Visits: Basal Visit (hospitalization), Visit at 3 days, Discharge Visit

SECONDARY OUTCOMES:
Effectiveness | 3 Visits: Basal Visit (hospitalization), Visit at 3 days, Discharge Visit

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A. (formerly Janssen Sp) Clinical Trial, Study Director — Janssen-Cilag, S.A.

REFERENCES:
- See also: Impact of aggressiveness/agitation in response and safety to risperidone in acute psychotic patients. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=281&filename=CR009214_CSR.pdf